CLINICAL TRIAL: NCT06992011
Title: A Randomized Controlled Trial Comparing Clinical Effectiveness of SMILE Versus SMILE Xtra in Myopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2024-267R-1
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMILE Group (Active Comparator)
  Interventions: Procedure: SMILE
- SMILE Xtra Group (Experimental)
  Interventions: Procedure: SMILE Xtra

INTERVENTIONS:
Procedure: SMILE — Small Incision Lenticule Extraction
  Arms: SMILE Group
Procedure: SMILE Xtra — Small Incision Lenticule Extraction combined with Corneal Cross-linking (SMILE Xtra)
  Arms: SMILE Xtra Group

SUMMARY:
To evaluate and compare the clinical efficacy, biomechanical stability, and optical quality of SMILE and SMILE Xtra procedures in patients with myopia through a randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years
2. MRSE (Manifest Refraction Spherical Equivalent) -6.00D to -10.00D with refractive changes within ±0.50D in past 2 years
3. CDVA (Corrected Distance Visual Acuity) ≥ 20/25
4. Myopia progression ≤ 0.50D/year for ≥2 years
5. RST (Residual Stromal Thickness) ≥ 250μm after lenticule removal
6. Contact lens discontinuation as per protocol

Exclusion Criteria:

1. Other eye diseases (keratoconus, glaucoma, etc.)
2. Corneal scarring, cataracts affecting observation
3. Systemic diseases affecting surgery compliance
4. Prior ocular surgeries
5. Pregnancy, breastfeeding, or menstruation
6. Drug allergies to surgical medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 1 week, 1 month,3 months， 6 months, 12 months, 24 months, and 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China